CLINICAL TRIAL: NCT01752127
Title: Study for Investigate the Effectiveness and Safety of Resolute Integrity or Xience Prime in Diabetes or Small Vessels Lesion Patients
Brief Title: COmparison of Xience PrimE Versus REsolute Integrity in Diabetes or Small Vessel Disease
Acronym: COPERES
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Lae Young Jung, Doctor, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The COPERES trial
Record Dates: First submitted 2012-12-02; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Angioplasty, Balloon, Coronary
Keywords: Drug-eluting stent; diabetes; small vessel disease
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- DM arms (Active Comparator): comparison of two different stents(Xience prime and Resolute integrity)
  Interventions: Procedure: percutaneous coronary intervention using drug eluting stent
- Small vessel arms (Active Comparator): comparison of two different stents(Xience prime and Resolute integrity)
  Interventions: Procedure: percutaneous coronary intervention using drug eluting stent

INTERVENTIONS:
Procedure: percutaneous coronary intervention using drug eluting stent — 1. Intracoronary stenting
  1. The procedure could be conducted via brachial, radial or femoral approaches.
  2. There are no restrictions regarding lesion's length or diameter. For long lesions, overlapping of several stents would be allowed but only allocated type of stents should be used.
  3. When several lesions are included in the study of a patient, each lesion may be allocated in different groups. Only if deployment of the allocated stent is not possible, crossing to other stent would be allowed.
  4. Direct stenting or bifurcation stenting is allowed.
  5. Predilation before stenting, IVUS examination, and administration of glycoprotein IIb/IIIa inhibitor would be determined by investigator.
  Other Names: using two drug eluting stent(XIENCE PRIME and RESOLUTE INTEGRITY)

SUMMARY:
The newer generation ZES (Medtronic, Minneapolis, MN, Resolute Integrity) and EES (Abbott Vascular, Abbott Park, Illinois, Xience Prime) were introduced to South Korea. Although these are thought to be superior in effect and stability compared to ZES and EES of previous generation, there are few clinical data regarding the high risk groups of diabetes patients or small vessels lesion. Moreover, looking at the 8.3% of restenosis in Resolute All Comer study (23% diabetes), the investigators could not know the outcome in high risk patients such as diabetes or small vessels lesion. Therefore, the aim of this study is to investigate the effectiveness and safety of Resolute Integrity or Xience Prime in diabetes or small vessels lesion patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Patients requiring stent procedure (visual diameter stenosis ≥ 50%)
3. Stable angina with evidence of myocardial ischemia, acute coronary syndrome(ST segment elevation, non-ST segment elevation acute myocardial infarction, and unstable angina)
4. Patients diagnosed of type 2 diabetes or small vessel disease
5. Patients willing to participate in the study through written consent

Exclusion Criteria:

1. Those hypersensitive to or abstaining from heparin, aspirin, clopidogrel, contrast medium, zotarolimus, or everolimus.
2. Pregnant women or those having future plans for pregnancy.
3. Those having hemorrhagic disease or blood-clotting disorders (including heparin-induced thrombocytopenia), or those rejecting blood transfusion.
4. Those having medical history of digestive and urinary system bleeding during the last 3 months, or who have received major surgery within 2 months.
5. Those with thrombocytopenia (< 100,000/mm3) or hemoglobin 10.0 g/dL or less.
6. Those planning a surgery that requires the discontinuation of antiplatelet drugs within next 12 months (especially, thienopyridines type).
7. When the remaining survival period is expected to be less than 1 year.
8. Restenosis lesion
9. Left main coronary artery lesion
10. Saphenous vein graft stenosis lesion
11. Left ventricular ejection fraction < 30%
12. Cardiac shock
13. Those with liver function failure: When liver enzyme level (ALT) is 3 times the normal upper limit.
14. Type I diabetes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
in-segment late lumen loss (mm)at 12month | 12month

SECONDARY OUTCOMES:
major adverse cardiac events(MACE) at 12month | 12month
  1) Occurrence of major adverse cardiac events (MACE) during 12 months
  * Cardiac death
  * Target vessel related myocardial infarction
  * Ischemia driven Target Vessel Revascularization (TVR)
  * Ischemia driven Target Lesion Revascularization (TLR)
  * Definite / probable stent thrombosis by ARC definition
MACE at 24month | 24month
  2) Occurrence of major adverse cardiac events (MACE) during 24 months
  * Cardiac death
  * Target vessel related myocardial infarction
  * Ischemia driven Target Vessel Revascularization (TVR)
  * Ischemia driven Target Lesion Revascularization (TLR)
  * Definite / probable stent thrombosis by ARC definition
procedure success rate | 1 day (after procedure)
  Procedure success rate proportion of investigational stent deployed successfully without chage to other stent

CONTACTS AND LOCATIONS:
Locations (1):
- Devision of cardiology, Chonbuk national university hospital, Jeonju, Chon-buk, South Korea